CLINICAL TRIAL: NCT02553005
Title: Evaluation of the Effect of Acupuncture on Hand Pain, Functional Deficits and Health Related Quality of Life in Patients With Rheumatoid Arthritis - A Multicenter, Double-blinded, Randomised Clinical Trial
Brief Title: Evaluation of the Effect of Acupuncture on Hand Pain, Functional Deficits and Health Related Quality of Life in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Susana Seca, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of Coimbra
Record Dates: First submitted 2015-09-12; First posted 2015-09-17 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Acupuncture
Keywords: Acupuncture; Rheumatoid Arthritis; Quality of life; Hand Strength
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- sham acupuncture (Sham Comparator): False acupuncture treatment using not acupuncture points
  Interventions: Procedure: Acupuncture
- verum acupuncture (Experimental): Real acupuncture treatment
  Interventions: Procedure: Acupuncture
- Control (No Intervention)

INTERVENTIONS:
Procedure: Acupuncture
  Arms: sham acupuncture; verum acupuncture

SUMMARY:
Rheumatoid Arthritis (RA) is a systemic inflammatory disease characterized by functional disability and pain. Although acupuncture is widely used, western acupuncture studies on RA show no conclusive positive result. Acupuncture is regarded as a reflex therapy, and Traditional Chinese Medicine (TCM) diagnosis was shown to be an individual neurovegetative state allowing to individually allocated acupoints. Positive results were reported using a classical diagnostic procedure to allocate acupoints to the patient according to the Shang Han Lun. The investigators are interested if acupuncture compatible with this ancient theory would be successful in improve hand function in RA patients.

The investigators therefore developed a prospective randomized control trial in a three-armed parallel group design with a standardized treatment intervention. Only patients with the TCM diagnosis of a so-called Turning Point syndrome will be allowed in the experimental phase. This may harmonize TCM diagnosis and the standardized intervention, in order to optimize potential therapeutic effects.

DETAILED DESCRIPTION:
The study design is divided into two parts. First the investigators will follow a non-experimental nature design. Based on the results of this exploratory study we will then start a three-armed parallel-group study with equal randomization (1:1:1), prospective, double-blind, placebo-controlled and multicenter that will be conducted in Portugal (2 sites).

We plan to include 381 patients with RA of the hands in accordance to the selection criteria. The patients are going to be recruited from the national centers of rheumatology and patient associations in the time from May 2015 to October 2016. All patients are supposed to sign an informed consent at the time of enrollment according to the rules of the Helsinki Declaration.

Task 1 In the first task we are going to develop a non-experimental, exploratory and descriptive nature design with the goal to describe the epidemiological, clinical and genetic profile of patients with RA of the hands according to their TCM diagnosis.

We will use an individual instrument for the collection of data to characterize the patients socio-demographically and clinically.

The main characteristics, complaints and objective examinations of participants, will be characterized by a qualified and experienced acupuncturist (first physician), in accordance to the Heidelberg Model (HM) to TCM. This physician will assess the pain in the hand by using a pressure algometer in two different distinct points. It is well known that the lower the ability to tolerate the pressure is, the worse will be the individual pain. The same researcher will also record clinical features based on data from tongue-diagnosis that will have been conducted before by an Automatic Tongue Diagnosis System (ATDS). The results so far demonstrate that the ATDS is very consistent even in settings with different environmental lighting.

The correlation between pattern classification in TCM and biomarkers that are expressed in genetic profiles in RA patients will be explored similarly to other recent studies whose results indicated that different patterns could be regarded as a consequence of biological networks with deviant gene expressions in various affected tissues and immune effector cells.

Due to financial limitations, we will only select 15 participants randomly from each of the different TCM patterns found. Eight ml of venous blood will be collected in anticoagulation tubes from each participant and will then be tested in a microarray assay by using the Trizol extraction method.

Task 2 Next, we aim to evaluate the effect of acupuncture on pain and strength of the hand according to the criteria of the HM to TCM for a specific vegetative functional state called the TP syndrome.

A sample of 90 patients with clinical features of a TP syndrome will be assigned randomly to one of three parallel groups, in a 1:1:1 ratio to either the control, verum or sham group with the help of a computer-generated randomization programme.

The first physician will mark the points with a red or blue colour on the patients that have been randomized to the verum intervention group as well as on the patients that have been assigned to the sham intervention group.

Afterwards, the first physician will present these data to a study-coordination program that will assign the colour-codes to a sequence of possible treatment modalities by using a computer-generated randomization table. A second physician will then be informed by the programme about the colour of the points that is supposed to be needled. The second physician will then perform a respective standardized needling technique to the selected points indicated by the colour which corresponds to either the sham or verum points.

We decided to use the Leopard Spot technique, a blood-letting acupuncture therapy that uses sterile subcutaneous needles (0,30mmx8mm) and it is known to increase local microcirculation by inducing a vegetative response. All patients will receive three sessions of treatment. After the acupuncture session, the patients must dress with light garment to cover any potential marks from needling.

Before and after the treatments, the patients will return to the first physician for the assessment of the outcomes. The first physician will not know which acupuncture points have been used.

The participants will be followed up for six times Assessment (0) will take place after randomization; assessments (1), (3) and (5) will take place five minutes after the intervention; assessment (2) will be done 24 hours after the first intervention and assessment (4) three days after the first intervention.

The assessments include an evaluation of the patients tolerance to pain in the hand by using a pressure algometer; a measurement of their grip strength with the help of a dynamometer and an evaluation of the nerve conduction and muscle function in the hand using an electromyography.

Task 3 In this task we intend to do a longitudinal study to assess the effect of the acupuncture treatment on inflammation and on the quality of life.

The patients that had been randomized to groups 2 and 3 will be treated two times per week, over a period of three weeks, respecting an interval of 72 hours in between treatments. Therefore these participants will be followed up in the assessments (6), (8), (10), (12), (14) and (16) - (before intervention) and assessments (7), (5), (9), (11), (13), (15) and (17) - (five minutes after intervention) (Appendix 6). The assessments (0), (5) and (18) will also include another parameter to measure the inflammation condition: the cortisol and interleukins level in the saliva.

All the patients randomized to groups 1, 2 and 3 will be followed up in the assessments (0) and (18) - 28 days after assessment (0), also to measure of pain by Visual Analogue Scale and of quality of life by Health Survey SF-36.

The results of the first task will be conducted by analyzing statistical data, using techniques of descriptive statistics and nonparametric tests. To the second and third tasks the results will be analyzed by Pearson Correlation Coefficients and a Multivariate Analysis of Variance with the significance set at p<0,05.

ELIGIBILITY:
Inclusion Criteria:

* Compliance inform consent
* Patients with RA
* Fulfill The ACR criteria of RA
* Impairment of the hand strength with or without pain in the hands during the grip procedure
* Chronic pain: either persistent or intermittent over a minimum period of three months prior to recruitment
* Current pain: greater than 30/ 100 mm on a pain visual analogue scale (VAS) within the last 24 hours despite medication
* Patients on stable dose treatment for at least 3 weeks

Exclusion Criteria:

* Under the age of 18 years
* Previously had acupuncture
* Localized skin infections
* Severe chronic or uncontrolled co-morbid disease
* The wish to get a pension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-10 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
gene expression profiles (Assessment by microarray) | up to 19 months
  Assessment by microarray
Quality of life (Assessment by SF-36 scale) | up to 19 months
  Assessment by SF-36 scale

SECONDARY OUTCOMES:
Cortisol levels in blood | up to 12 months
  Assessment by cortisol levels in blood
Interleucines levels in blood | up to 12 months
  Assessment by interleucines levels in blood
hand pain (Assessment by algometry) | up to 19 months
  Assessment by algometry
hand strength (Assessment by dynamometry) | up to 19 months
  Assessment by dynamometry

CONTACTS AND LOCATIONS:
Overall Officials: Susana Seca, MSc, Principal Investigator — University of Coimbra
Locations (1):
- Faculty of Medicine - University of Coimbra, Coimbra, Coimbra District, Portugal

REFERENCES:
- [Derived] Seca S, Kirch S, Cabrita AS, Greten HJ. Evaluation of the effect of acupuncture on hand pain, functional deficits and health-related quality of life in patients with rheumatoid arthritis--A study protocol for a multicenter, double-blind, randomized clinical trial. J Integr Med. 2016 May;14(3):219-27. doi: 10.1016/S2095-4964(16)60254-6. PMID 27181129